CLINICAL TRIAL: NCT06497270
Title: A 3D Bioprinted Hormone-producing Model for BRCA Mutated Patients After Risk Reducing Surgery: the DISC-OVARY Trial
Acronym: DISC-OVARY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, MARCHETTI CLAUDIA, Professor, MD PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DISC-OVARY
Record Dates: First submitted 2024-06-26; First posted 2024-07-11 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: BRCA Mutation; Estrogen Deficiency; Surgical Menopause; Menopause Related Conditions; Menopause, Premature; Ovarian Cancer
Keywords: BRCA mutation; Surgical menopause; ovarian cancer prevention; estrogen deficiency
MeSH Terms: conditions — Menopause, Premature; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: PILOT study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRCAmut patients (Experimental): germinal BRCA1/2 mutated (BRCAmut) patients undergoing risk reducing salpingo-oophorectomy whose ovaries will be used to select theca and granulosa cells for the 3D bioprinted device.
  Interventions: Procedure: Theca and Granulosa Cell Isolation

INTERVENTIONS:
Procedure: Theca and Granulosa Cell Isolation — These patients will receive standard procedure during the risk reducing surgery but their ovaries will be used to extract theca and granulosa cells which will be used for the 3D bioprinted device's realisation.

SUMMARY:
Selecting theca and granulosa cells from removed ovaries of BRCA1/2mut patients undergoing Risk-reducing salpingo-oophorectomy (RRSO) and developing a 3D bioprinted hormone-producing bioprosthetic model. If efficacy and tolerability are confirmed in vivo, this bioprosthetic model might be used to replace hormones' production in BRCA mutated patients undergoing prophylactic surgery.

DETAILED DESCRIPTION:
Background and Rationale Women carrying germline BReast CAncer gene (BRCA) 1/2 mutations have an increased lifetime risk of breast and ovarian cancers (72% and 44% for BRCA1 and 69% and 17% for BRCA2, respectively). Risk-reducing salpingo-oophorectomy (RRSO) by the age of 40 (postponable to age of 45 for BRCA2mut) is the standard of care in ovarian cancer risk reduction (about 80%). Although potentially lifesaving, RRSO may negatively affect quality of life and impair long-term health (cardiovascular disease, osteoporosis and impairment of immune response).

To overcome these side effects, hormone replacement therapy (HRT) is crucial but remains a major concern, especially due to its negative effects (potential breast cancer risk, thromboembolic events) and, overall, due to the long-term safety lack of data. Synthetic and animal-derived hormones seem to be associated with breast cancer risk. Although breast cancer risk is lower for bioidentical hormones (i.e. estriol), data continue to be discordant. Several evidence still sustain estriol's impact on breast cancer (especially for lobular histotype; OR 2.0, 95% CI 1.3-3.2) and endometrial disease (endometrial cancer: OR 3.0, 95% CI 2.0-4.4 and endometrial atypical hyperplasia: OR 8.3, 95% CI 4.0-17.4, respectively). Furthermore, estriol's efficacy on cardiovascular disease and osteoporosis is still unclear when compared to other estrogen compounds. Side effects of estriol therapy may include breast tenderness, nausea, bloating, mood changes, headache, and vaginal bleeding or spotting. Moreover, all the HRT's administration routes (oral, transdermal, and vaginal) need daily/frequent assumption, thus compliance of the patients is essential and adherence to long-term therapy in developed countries is reported around 50% with a high risk of forgetfulness or discontinuation. Each route also has specific disadvantages (i.e. the risk of thromboembolism in the oral one). Finally, HRT may influence other hormones' production: it increases T4 dosage requirements of women being treated for primary hypothyroidism as well as alter the pituitary-thyroid axis in euthyroid women. While for cortisol level findings are still inconsistent, hormone exogenous intake does not permit to follow the daily hormonal fluctuation. Aging and hypoestrogenism, in postmenopausal women, determine immune system changes which may play a crucial role in the development of postmenopausal diseases (diabetes or atherosclerosis) and may be negatively influenced by HRT. Preliminary data of a recent MITO group survey revealed that only 70% of gynecologists recommend HRT after RRSO due to oncological safety concerns and low women's requests (more than 70% of cases were oral prescriptions, while only 24% preferred local administration).

In conclusion, for some women, the concern of menopause risks act as a deterrent for a lifesaving procedure (RRSO). In this scenario, it is fundamental to provide a new strategy for BRCA mutated patients, in order to reduce menopausal drawbacks without exposing participants to a higher breast cancer risk, reproducing the physiological hormonal rhythm without compliance issue. The 3D bioprinted hormone-producing model from patients' own autologous cells could meet this need.

HYPOTHESIS The investigators hypothesize to select theca and granulosa cells from removed ovaries of BRCA1/2mut patients undergoing RRSO, avoiding the epithelial ones at risk of developing cancer, and use those cells to develop a 3D bioprinted hormone-producing bioprosthetic model in order to replace patients' own production.

AIMS Primary endpoint: Restore normal estrogen and progesterone serum level in participants undergoing RRSO by the 3D bioprinted hormone-producing model's implant.

EXPERIMENTAL DESIGN No study has previously investigated the feasibility of 3D bioprinted hormone-producing model, hence this configures as a pilot study which, as such, does not need any formal sample size calculation.

The proposed research project aims to select theca and granulosa cells from patients' removed ovaries, combine them with different ratios of extracted mesenchymal cells; print them onto the prosthetic model scaffolds and assess the hormone production.

IMPACT ON CANCER The results of the pilot project will provide a 3D bioprinted model able to produce estrogens and progesterone in vitro. If functionality is confirmed in vivo, the model might be used in BRCA mutated patients allowing them to avoid surgery induced menopause's side effects. Specifically, a 3D bioprinted hormone-producing bioprosthetic model would provide patients with a viable alternative to surgery-induced menopause and traditional HRT.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18-40 years old;
* BRCA1/2 germline mutations;
* Completed childbearing;
* Willing to undergo RRSO;
* Negative final histological examination;
* No previous breast cancer.

Exclusion Criteria:

* Other malignancies;
* Final histological examination reporting malignant disease (any);
* Desire of fertility sparing.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 3 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
oestrogens and progesterone's levels | minumum 3 months
  (Unit: pg/mL for both hormones)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Marchetti, Professor, Principal Investigator — Policlinico Universitario Fondazione Agostino Gemelli, IRCCS, Rome, Italy
Locations (1):
- Day Hospital Tumori Femminili, Policlinico Universitario Fondazione Agostino Gemelli, IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antoniou A, Pharoah PD, Narod S, Risch HA, Eyfjord JE, Hopper JL, Loman N, Olsson H, Johannsson O, Borg A, Pasini B, Radice P, Manoukian S, Eccles DM, Tang N, Olah E, Anton-Culver H, Warner E, Lubinski J, Gronwald J, Gorski B, Tulinius H, Thorlacius S, Eerola H, Nevanlinna H, Syrjakoski K, Kallioniemi OP, Thompson D, Evans C, Peto J, Lalloo F, Evans DG, Easton DF. Average risks of breast and ovarian cancer associated with BRCA1 or BRCA2 mutations detected in case Series unselected for family history: a combined analysis of 22 studies. Am J Hum Genet. 2003 May;72(5):1117-30. doi: 10.1086/375033. Epub 2003 Apr 3. PMID 12677558
- [Background] Gabaldo Barrios X, Sarabia Meseguer MD, Marin Vera M, Sanchez Bermudez AI, Macias Cerrolaza JA, Sanchez Henarejos P, Zafra Poves M, Garcia Hernandez MR, Cuevas Tortosa E, Aliaga Bano A, Castillo Guardiola V, Martinez Hernandez P, Tovar Zapata I, Martinez Barba E, Ayala de la Pena F, Alonso Romero JL, Noguera Velasco JA, Ruiz Espejo F. Molecular characterization and clinical interpretation of BRCA1/BRCA2 variants in families from Murcia (south-eastern Spain) with hereditary breast and ovarian cancer: clinical-pathological features in BRCA carriers and non-carriers. Fam Cancer. 2017 Oct;16(4):477-489. doi: 10.1007/s10689-017-9985-x. PMID 28477318
- [Background] Marchetti C, De Felice F, Palaia I, Perniola G, Musella A, Musio D, Muzii L, Tombolini V, Panici PB. Risk-reducing salpingo-oophorectomy: a meta-analysis on impact on ovarian cancer risk and all cause mortality in BRCA 1 and BRCA 2 mutation carriers. BMC Womens Health. 2014 Dec 12;14:150. doi: 10.1186/s12905-014-0150-5. PMID 25494812
- [Background] Rocca WA, Grossardt BR, de Andrade M, Malkasian GD, Melton LJ 3rd. Survival patterns after oophorectomy in premenopausal women: a population-based cohort study. Lancet Oncol. 2006 Oct;7(10):821-8. doi: 10.1016/S1470-2045(06)70869-5. PMID 17012044
- [Background] Madalinska JB, Hollenstein J, Bleiker E, van Beurden M, Valdimarsdottir HB, Massuger LF, Gaarenstroom KN, Mourits MJ, Verheijen RH, van Dorst EB, van der Putten H, van der Velden K, Boonstra H, Aaronson NK. Quality-of-life effects of prophylactic salpingo-oophorectomy versus gynecologic screening among women at increased risk of hereditary ovarian cancer. J Clin Oncol. 2005 Oct 1;23(28):6890-8. doi: 10.1200/JCO.2005.02.626. Epub 2005 Aug 29. PMID 16129845
- [Background] Gaba F, Blyuss O, Chandrasekaran D, Osman M, Goyal S, Gan C, Izatt L, Tripathi V, Esteban I, McNicol L, Ragupathy K, Crawford R, Evans DG, Legood R, Menon U, Manchanda R. Attitudes towards risk-reducing early salpingectomy with delayed oophorectomy for ovarian cancer prevention: a cohort study. BJOG. 2021 Mar;128(4):714-726. doi: 10.1111/1471-0528.16424. Epub 2020 Aug 16. PMID 32803845
- [Background] Kumru S, Godekmerdan A, Yilmaz B. Immune effects of surgical menopause and estrogen replacement therapy in peri-menopausal women. J Reprod Immunol. 2004 Aug;63(1):31-8. doi: 10.1016/j.jri.2004.02.001. PMID 15284002
- [Background] Rott H. Prevention and treatment of venous thromboembolism during HRT: current perspectives. Int J Gen Med. 2014 Sep 1;7:433-40. doi: 10.2147/IJGM.S46310. eCollection 2014. PMID 25210472
- [Background] Bakken K, Alsaker E, Eggen AE, Lund E. Hormone replacement therapy and incidence of hormone-dependent cancers in the Norwegian Women and Cancer study. Int J Cancer. 2004 Oct 20;112(1):130-4. doi: 10.1002/ijc.20389. PMID 15305384
- [Background] Holtorf K. The bioidentical hormone debate: are bioidentical hormones (estradiol, estriol, and progesterone) safer or more efficacious than commonly used synthetic versions in hormone replacement therapy? Postgrad Med. 2009 Jan;121(1):73-85. doi: 10.3810/pgm.2009.01.1949. PMID 19179815
- [Background] Rosenberg LU, Magnusson C, Lindstrom E, Wedren S, Hall P, Dickman PW. Menopausal hormone therapy and other breast cancer risk factors in relation to the risk of different histological subtypes of breast cancer: a case-control study. Breast Cancer Res. 2006;8(1):R11. doi: 10.1186/bcr1378. Epub 2006 Feb 17. PMID 16507159
- [Background] Weiderpass E, Baron JA, Adami HO, Magnusson C, Lindgren A, Bergstrom R, Correia N, Persson I. Low-potency oestrogen and risk of endometrial cancer: a case-control study. Lancet. 1999 May 29;353(9167):1824-8. doi: 10.1016/S0140-6736(98)10233-7. PMID 10359406
- [Background] Furness S, Roberts H, Marjoribanks J, Lethaby A. Hormone therapy in postmenopausal women and risk of endometrial hyperplasia. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD000402. doi: 10.1002/14651858.CD000402.pub4. PMID 22895916
- [Background] Faulkner DL, Young C, Hutchins D, McCollam JS. Patient noncompliance with hormone replacement therapy: a nationwide estimate using a large prescription claims database. Menopause. 1998 Winter;5(4):226-9. PMID 9872489
- [Background] Skouby SO, Barlow D, Samsioe G, Gompel A, Pines A, Al-Azzawi F, Graziottin A, Hudita D, Rozenberg S; European Menopause and Andropause Society (EMAS). Climacteric medicine: European Menopause and Andropause Society (EMAS) statements on postmenopausal hormonal therapy. Maturitas. 2004 May 28;48(1):19-25. doi: 10.1016/j.maturitas.2004.03.003. PMID 15223104
- [Background] Lumsden MA. The NICE Guideline - Menopause: diagnosis and management. Climacteric. 2016 Oct;19(5):426-9. doi: 10.1080/13697137.2016.1222483. Epub 2016 Aug 24. No abstract available. PMID 27558301
- [Background] Mazer NA. Interaction of estrogen therapy and thyroid hormone replacement in postmenopausal women. Thyroid. 2004;14 Suppl 1:S27-34. doi: 10.1089/105072504323024561. PMID 15142374
- [Background] Edwards KM, Mills PJ. Effects of estrogen versus estrogen and progesterone on cortisol and interleukin-6. Maturitas. 2008 Dec 20;61(4):330-3. doi: 10.1016/j.maturitas.2008.09.024. Epub 2008 Nov 17. PMID 19010617
- [Background] Abdi F, Mobedi H, Roozbeh N. Hops for Menopausal Vasomotor Symptoms: Mechanisms of Action. J Menopausal Med. 2016 Aug;22(2):62-4. doi: 10.6118/jmm.2016.22.2.62. Epub 2016 Aug 30. PMID 27617238
- [Background] Taneja V. Sex Hormones Determine Immune Response. Front Immunol. 2018 Aug 27;9:1931. doi: 10.3389/fimmu.2018.01931. eCollection 2018. No abstract available. PMID 30210492
- [Background] Gradishar WJ, Moran MS, Abraham J, Abramson V, Aft R, Agnese D, Allison KH, Anderson B, Burstein HJ, Chew H, Dang C, Elias AD, Giordano SH, Goetz MP, Goldstein LJ, Hurvitz SA, Jankowitz RC, Javid SH, Krishnamurthy J, Leitch AM, Lyons J, Mortimer J, Patel SA, Pierce LJ, Rosenberger LH, Rugo HS, Schneider B, Smith ML, Soliman H, Stringer-Reasor EM, Telli ML, Wei M, Wisinski KB, Young JS, Yeung K, Dwyer MA, Kumar R. NCCN Guidelines(R) Insights: Breast Cancer, Version 4.2023. J Natl Compr Canc Netw. 2023 Jun;21(6):594-608. doi: 10.6004/jnccn.2023.0031. PMID 37308117

DOCUMENTS (1):
  • Study Protocol (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT06497270/Prot_000.pdf